CLINICAL TRIAL: NCT07185789
Title: Multidimensional Intervention to Improve Healthy Lifestyle Practices and Nutrition and Health Status in Mexican Schoolchildren: Development of an Intervention Platform, Randomized Clinical Trial and Scaling Proposal
Brief Title: Multidimensional Intervention in Mexican Schoolchildren
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican National Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Edgar Denova Gutierrez, Principal Investigator, Mexican National Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MexicanNIPH
Record Dates: First submitted 2024-04-07; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Childhood Obesity; Pediatric Obesity; Childhood Overweight
Keywords: Childhood obesity; School children
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: The children who participate are not aware of being a control or intervention group, as well as their parents, teachers and school cooperative staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervención Multidimensional (Active Comparator): The multidimensional intervention will be received in 10 schools in 3 states of Mexico (Campeche, Mexico City and Morelos). In these schools, an initial diagnosis of the environment, monitoring and evaluation of the implemented strategies will be carried out. Subsequently, a baseline measurement will be carried out, where anthropometric, behavioral and environmental modification indicators will be evaluated, including the measurement of body composition through dual x-ray absorption densitometry (DXA), cardiometabolic health indicators such as glycated hemoglobin (HbA1c), lipid profile, liver function and biological markers; inflammation markers. The intervention will include activities related to: A) Healthy and sustainable eating; B) Movement behaviors; C) Psychosocial determinants. Finally, a final measurement will be carried out where the same variables as in the initial measurement will be evaluated.
  Interventions: Behavioral: Healthy and Sustainable Eating; Behavioral: Movement behaviors; Behavioral: Psychosocial determinants
- Control (No Intervention): Multidimensional intervention will not be received. In these schools, an initial diagnosis of the environment will be carried out, monitoring and evaluation of the strategies implemented and a more in-depth initial and basal measurement will be carried out, using anthropometric, behavioral and environmental modification indicators, including the measurement of body composition through dual x-ray absorption densitometry (DXA), cardiometabolic health indicators such as glycated hemoglobin (HbA1c), lipid profile, liver function and biological markers; inflammation markers.
  A final measurement will be carried out to compare the results.

INTERVENTIONS:
Behavioral: Healthy and Sustainable Eating — Animated projections, snacks that incorporate fruits and/or vegetables, measuring their hydration status through images where they can observe the color of their urine and relate it to the amount of plain water they have consumed, as well as activities through the mobile messaging platform, WhatsApp.
  Other Names: Movement behaviors; Psychosocial determinants
  Arms: Intervención Multidimensional
Behavioral: Movement behaviors — Animated projections, snacks that incorporate fruits and/or vegetables, measuring their hydration status through images where they can observe the color of their urine and relate it to the amount of plain water they have consumed, as well as activities through the mobile messaging platform, WhatsApp.
  Arms: Intervención Multidimensional
Behavioral: Psychosocial determinants — Workshops on key topics of psychosocial determinants in children, virtual workshops on topics of psychosocial determinants such as obesity and healthy eating.
  Arms: Intervención Multidimensional

SUMMARY:
The aims is to evaluate the effects of an multidimensional intervention on the physical-built and social environment around schools and the nutritional status of the school population, through a randomized community trial, in schools in 3 states of the Mexican Republic, using anthropometric indicators, biological, psychological, behavioral and environmental.

The main questions it aims to answer are:

1. What are the main risk and protective factors for overweight and obesity in the school environment and in the environments around schools in primary education schools in three states of the Mexican Republic?
2. Is there a relationship between risky eating behaviors and the body mass index of schoolchildren?
3. Are the strategies that are being implemented effective in reducing the presence of risk factors and increasing the presence of protective factors for overweight and obesity in the school environment and in the environments around schools?
4. Are the strategies that are being implemented effective in reducing the presence of risk factors and increasing the protective factors for overweight and obesity in the family environment?

DETAILED DESCRIPTION:
This is a project designed and approved to be carried out in 4 stages. The project has financing from the health sector fund and also an extension to end on January 11, 2025. The objective is to evaluate the effects of a multidimensional intervention (MI) on the physical-built and social environment around schools, as well as, on the nutritional status of the school population, through a community trial in schools in 3 states of the Mexican Republic (Campeche, Mexico City and Morelos). The impact will be measured through anthropometric, biological, psychological, behavioral and environmental indicators. The target population of the intervention will be students between 9-12 years old who are in the 4th grade of primary school.

Stage 1. Situational diagnosis. Duration: 12 months. In the design of health promotion interventions, situational diagnostic assessment is necessary to be able to design an intervention adapted to the context and real needs of the target population. This stage of the project also allows us to identify previous experiences and derive from them available evidence on interventions that have been implemented in other populations. Likewise, it is necessary to identify the health problems of the population to which the intervention to be designed is directed, as well as the existing policies and programs and the participation of the target population to which the intervention to be designed is aimed.

Stage 2. Design and development of the multidimensional intervention and evaluation instruments. Duration: 12 months. The information generated from the situational diagnosis will serve to design the multidimensional intervention of this proposal, which will include different levels of intervention such as school, around school, home and community. The components of this stage are the following: 1) Final design of the multidimensional intervention; and 2) Definition of the components of the multidimensional intervention, which include: a) Actions to ensure a healthy food environment; b) Comprehensive Physical Activity Program; c) Teacher training; d) Motivation of teachers; e) Educational materials with a social marketing focus, short or simple message service (SMS), printed or audiovisual material; f) Implementation logistics; g) Development of instruments necessary for intervention; h) Validation or pilot testing of the intervention materials.

Stage 3. Implementation, monitoring and evaluation of the multidimensional intervention. Duration: 10 months. The final design of the multidimensional intervention that will be implemented during this stage will depend on the modifications made in the stages described above. This stage consists of the following phases: 1) Randomization, 2) Initial evaluation, 3) Beginning of the intervention, 4) Monitoring and evaluation of the process and 5) Final evaluation.

Stage 4. Institutionalization of the intervention. Duration: 12 months. In the final stage, an analysis and formulation of recommendations will be carried out for the escalation and incorporation of the intervention to the Ministry of Public Education (SEP, for its acronym in Spanish).

The study consists of a community trial in 24 schools in 3 states of the Mexican Republic (Campeche, Morelos and Mexico City) and a parallel randomized clinical trial in 4 of the schools in Cuernavaca, Morelos. Both studies together will address the questions raised in the previous section.

ELIGIBILITY:
Inclusion Criteria:

* Fourth grade elementary schools children from schools that belong to Federal entities: Campeche, Morelos and Mexico City, with morning schedule, from 8:00 to 12:30 or extended schedule, from 8:00 to 14:00hrs.
* For Morelos State, elementary schools will be sought to be private, with at least 1000 enrollement students, with morning schedule, from 8:00 to 12:30 or extended schedule, from 8:00 to 14:00hrs.

Exclusion Criteria:

* Children that don´t correspond to the selected shifts.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — girls and boys have similiar proportion
Enrollment: 200 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic and Lipid Profile | Baseline and after 6 moths
  This outcome is designed to provide a fundamental assessment of the participant's cardiometabolic health status at the beginning of the study. It focuses on measuring key circulating molecules that are central to energy metabolism and cardiovascular risk.
  To achieve this, we will collect blood samples and analyze them for the core analytes that constitute a standard lipid panel and metabolic check:
  Glucose (mg/dL) Total Cholesterol (mg/dL) HDL-c (%) Triglycerides (mg/dL)
  The concentration of each of these analytes will be determined using Enzymatic Spectrophotometry.
Markers of Inflammation | Baseline and after 6 months
  We will measure the levels of Leptin, Adiponectin, IL-6, Galectin-3, HbA1c. We ELISA for the proteins, HPLC for HbA1c.
  Units: The results for the proteins will be reported in ng/mL, HbA1c as a percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Barquera Cervera, PhD, Study Director — National Institute of public Health
Locations (1):
- Instituto Nacional de Salud Pública, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No
Confidential information

REFERENCES:
- [Background] Bonvecchio A, Safdie M, Monterrubio EA, Gust T, Villalpando S, Rivera JA. Overweight and obesity trends in Mexican children 2 to 18 years of age from 1988 to 2006. Salud Publica Mex. 2009;51 Suppl 4:S586-94. doi: 10.1590/s0036-36342009001000013. PMID 20464234
- [Background] Barquera S, Campos I, Rivera JA. Mexico attempts to tackle obesity: the process, results, push backs and future challenges. Obes Rev. 2013 Nov;14 Suppl 2:69-78. doi: 10.1111/obr.12096. PMID 24103026
- [Background] Rivera JA, Irizarry LM, Gonzalez-de Cossio T. Overview of the nutritional status of the Mexican population in the last two decades. Salud Publica Mex. 2009;51 Suppl 4:S645-56. doi: 10.1590/s0036-36342009001000020. No abstract available. PMID 20464241
- [Background] Hernandez-Cordero S, Cuevas-Nasu L, Moran-Ruan MC, Mendez-Gomez Humaran I, Avila-Arcos MA, Rivera-Dommarco JA. Overweight and obesity in Mexican children and adolescents during the last 25 years. Nutr Diabetes. 2017 Mar 13;7(3):e247. doi: 10.1038/nutd.2016.52. PMID 28287630
- [Background] Incledon E, Wake M, Hay M. Psychological predictors of adiposity: systematic review of longitudinal studies. Int J Pediatr Obes. 2011 Jun;6(2-2):e1-11. doi: 10.3109/17477166.2010.549491. Epub 2011 Jan 19. PMID 21247271
- [Background] O'Dea JA, Caputi P. Association between socioeconomic status, weight, age and gender, and the body image and weight control practices of 6- to 19-year-old children and adolescents. Health Educ Res. 2001 Oct;16(5):521-32. doi: 10.1093/her/16.5.521. PMID 11675800
- [Background] Palma-Coca O, Hernandez-Serrato MI, Villalobos-Hernandez A, Unikel-Santoncini C, Olaiz-Fernandez G, Bojorquez-Chapela I. Association of socioeconomic status, problem behaviors, and disordered eating in Mexican adolescents: results of the Mexican National Health and Nutrition Survey 2006. J Adolesc Health. 2011 Oct;49(4):400-6. doi: 10.1016/j.jadohealth.2011.01.019. Epub 2011 May 20. PMID 21939871

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT07185789/Prot_SAP_ICF_000.pdf